CLINICAL TRIAL: NCT05771584
Title: A Phase 2 Study to Evaluate the Safety and Immunological Efficacy of Therapeutic Cancer Vaccine (AST-301, pNGVL3-hICD) in Patients With HER2 Expressing Gastric Cancer (CORNERSTONE-003)
Brief Title: Therapeutic Cancer Vaccine (AST-301, pNGVL3-hICD) in Gastric Cancer
Acronym: Conerstone3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aston Sci. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PN-301-22
Record Dates: First submitted 2022-09-06; First posted 2023-03-16 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sargramostim

STUDY DESIGN:
Intervention Model Description: Phase 2, open label, randomized, early proof-of-concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Total 300 μg of AST-301 (Experimental): AST-301/rhuGM-CSF (3-week interval, 3 cycles in total)
  Interventions: Drug: AST-301; Drug: rhuGM-CSF
- Total 600 μg of AST-301 (Experimental): AST-301/rhuGM-CSF (3-week interval, 6 cycles in total)
  Interventions: Drug: AST-301; Drug: rhuGM-CSF

INTERVENTIONS:
Drug: AST-301 — 100 μg
  Other Names: pNGVL3-hICD
Drug: rhuGM-CSF — 100 μg
  Other Names: Leukine; Sargramostim

SUMMARY:
The purpose of this early proof-of-concept study to evaluate the safety and immunologic efficacy of AST-301 in gastric cancer patients with HER2 expression (including both HER2 low expression and overexpression) who have completed the standard adjuvant treatment (including those who discontinued the standard adjuvant treatment due to intolerance).

Participants will be randomized 1:1 to either Arm 1 (Q3W, 3 cycles), or Arm 2 (Q3W, 6 cycles) of the study.

Safety Monitoring Committee (SMC) will oversee safety of study at 25% (6 participants), 50% (12 participants), and 75% (18 participants) of participants receive at least 1 dose of AST-301 and survival follow up will be performed to determine disease-free survival (DFS).

DETAILED DESCRIPTION:
Participants will provide informed consent and will undergo Pre-Screening/Screening procedures before taking part in the study. Participants will be in Arm 1 and Arm 2 will be conducted in parallel. AST-301 will be administrated every 3 weeks for a total of 3 immunizations in Arm 1 and a total of 6 immunizations in Arm 2.

* Arm 1: 3 immunizations of AST-301 admixed with immunoadjuvant recombinant human granulocyte-macrophage colony stimulating factor (rhuGM-CSF) administered at 3-week intervals. (Total 300 μg of AST-301)
* Arm 2: 6 immunizations of AST-301 admixed with immunoadjuvant recombinant human granulocyte-macrophage colony stimulating factor (rhuGM-CSF) administered at 3-week intervals. (Total 600 μg of AST-301) Randomization will be stratified according to HER2 expression (HER2 low expression or HER2 overexpression).

For both Arm 1 and Arm 2 of the study there will be a Pre-screen period, followed by study periods: a Screening Period (Day -28 to Day -1), a Treatment Period (3 cycles/Arm 1 and 6 cycles/Arm 2), an end of treatment (EOT) visit and follow-up visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Underwent a curative surgery with standard lymph node dissection (confirmed with no residual tumor, R0 resection) and have completed standard adjuvant treatment
* Has stages II or III according to the 8th edition of the American Joint Committee on Cancer (AJCC)
* HER2 low expression and HER2 overexpression diagnosed according to the 2016 College of American Pathologists (CAP)/American Society for Clinical Pathology (ASCP)/American Society of Clinical Oncology (ASCO) guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Demonstrates adequate organ function.

Key Exclusion Criteria:

* Has a history of hypersensitivity or other contraindications to rhuGM-CSF
* Has a history of other malignancies ≤5 years prior to first administration of Investigational Product (IP) except for adequately treated non-melanoma skin cancer or epithelial carcinoma without evidence of disease.
* Has received systemic immunosuppressants or were treated with systemic immunosuppressants ≤4 weeks prior to the first administration of Investigational Product (IP).
* Has a history of autoimmune disease or inflammatory disease
* Has active infection including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Is pregnant or breastfeeding or expecting to conceive children

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0. | up to 20 weeks
  To assess the safety of AST-301 administered in gastric cancer patients.
Immunologic efficacy of AST-301 immunization | 52 weeks
  AST-301 specific interferon (IFN)-gamma enzyme-linked immune absorbent spot (ELISpot) assay

SECONDARY OUTCOMES:
1year Disease-Free Survival rate (DFS rate) | 12 months
  disease free survival rate at 1 year
Disease-Free Survival rate (DFS rate) at end of study (EOS) | Overall study period approximately 31 months
  disease free survival at end of study
Compare immunogenicity of AST-301 between Arm 1 and Arm 2 | 52 weeks
  AST-301-specific IFN γ response by ELISpot assay
Change in central memory T-cell populations between Arm 1 and Arm 2 | 52 weeks
  Central memory T-cell (cluster of differentiation 4 (CD4) + and cluster of differentiation 8 (CD8) +) by a flow cytometry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hun Jung, MD, Study Director — jhun@astonsci.com
Locations (6):
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No